CLINICAL TRIAL: NCT00351182
Title: Phase 3 Study of Controlled Trial: 5-day Course of Telithromycin Versus Doxycycline for the Treatment of Mild to Moderate Scrub Typhus
Brief Title: Controlled Trial: 5-day Course of Telithromycin Versus Doxycycline for the Treatment of Mild to Moderate Scrub Typhus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-Min Kim (Other)
Responsible Party: Sponsor-Investigator, Dong-Min Kim, Chosun University Hospital, Chosun University Hospital
Organization: Chosun University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Telit_L_00276
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Scrub Typhus
Keywords: Scrub typhus; Telithromycin; Doxycycline
MeSH Terms: conditions — Scrub Typhus | interventions — telithromycin; Doxycycline

INTERVENTIONS:
Drug: Telithromycin
Drug: Doxycycline

SUMMARY:
New antibiotics are required that have antibacterial activity against doxycyline resistant O. tsutsugamushi, that can be safely used in pregnant women and children, that have a low possibility of inducing resistance and that do not induce cross resistant to other antibiotics. Telithromycin has been reported to be effective on Rickettsia, Batonella and Coxiella burnetii. Therefore, telithromycin may be considered as a substitute antibiotic that can be used safely in pregnant women and children for rickettsiosis or Orientia infection. Our study was designed to prove the clinical usefulness of telithromycin by comparing it with doxycycline for treating mild or moderate scrub typhus.

DETAILED DESCRIPTION:
Randomization and treatment assignment. After submitting a written, informed consent, the patients with an temperature of higher than 37.5°C and who met the eligibility criteria were randomly allocated to receive one of two oral regimens in accordance with a protocol that was determined by the last digit of a resident registration number (the patients with an odd number were treated by a5-daycourseofdaily 200-mg doses of doxycycline,and the patients with an even number were treated by a 5-day course of daily 800-mg doses of telithromycin). Therapy was started immediately after acomprehensive clinical examinationand the collection of specimens for laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

We conducted a multicenter prospective study of patients with possible scrub typhus. Adult patients (aged ≥18 years) who have had fever (temperature: ≥37.5°C) together with eschar or a maculopapular skin rash and ≥2 of the following symptoms: headache, malaise, myalgia, coughing, nausea, and abdominal discomfort, were enrolled after obtaining an informed consent from the patients or their guardians (10). Each patient was admitted between September, 2005 to December, 2005 to Chosun University Hospital or one of its two community branch hospitals (Jangheung Hospital and Chumdan Hospital), which are all located in southwest Korea.

Exclusion Criteria:

* The exclusion criteria were an inability to take oral medications, pregnancy, hypersensitivity to the trial drugs, previous drug therapy with potential antirickettsial activity (e.g., rifampicin, chloramphenicol, macrolides, fluoroquinolones or tetracyclines) within 48 h prior to admission, severe scrub typhus (shock requiring vasopressor therapy for >1 h, a stuporous or comatose level of consciousness, respiratory failure requiring mechanical ventilation or renal failure requiring immediate dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome was the fever clearance time; this was defined as the interval between the time at which the first dose of antibiotic was administered and the time at which the oral temperature first fell below 37.3°C and then it remained be

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Min Kim, Study Chair — Department of Internal Medidine, Chosun University Hospital
Locations (1):
- Chosun University Hospital, Gwangju, Jeollanam-do, South Korea